CLINICAL TRIAL: NCT04765865
Title: Evaluating Implementation and Scale-Up of Nigeria's National Sodium Reduction Program
Acronym: NaSS
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Abuja Teaching Hospital (Other); The George Institute (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Mark Huffman, Co-Director, Global Health Center; Professor of Medicine, Washington University School of Medicine
Other Study IDs: UATH/HREC/PR/2020/001; UG3HL152381 (NIH); UH3HL152381 (NIH)
Record Dates: First submitted 2021-02-18; First posted 2021-02-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Dietary Sources of Sodium; Population Sodium Intake
Keywords: Dietary Sodium; Sodium Intake; Sodium Reduction Program

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Wave 1: Participants will be enrolled as a single adult household representative from 3 states (Federal Capital Territory, Kano, Ogun) of Nigeria to complete a STEPs survey, 24-hour and spot urine assessments, blood sample collection for fatty acid estimation, and four (4) 24-hour dietary recalls (n=450).
  Interventions: Other: SHAKE Package
- Wave 2: Participants will be enrolled as a single adult household representative from 3 states (Federal Capital Territory, Kano, Ogun) of Nigeria to complete a STEPs survey and 24-hour and spot urine assessments (n=450).
  Interventions: Other: SHAKE Package
- Wave 3: Participants will be enrolled as a single adult household representative from 3 states (Federal Capital Territory, Kano, Ogun) of Nigeria to complete a STEPs survey, 24-hour and spot urine assessments, and four (4) 24-hour dietary recalls (n=450).
  Interventions: Other: SHAKE Package

INTERVENTIONS:
Other: SHAKE Package — The SHAKE (Surveillance of salt intake, Harness industry, Adopt standards for labelling and marketing, Knowledge to empower consumers, and Environments to promote health eating) package is a WHO Best Buy and is recently implemented within Nigeria by the Nigerian Agency for Food and Drug Administration and Control (NAFDAC).

SUMMARY:
The NaSS aims to assess the extent to which the SHAKE program is implemented within Nigeria by the Nigerian Agency for Food and Drug Administration and Control (NAFDAC) using a type III hybrid, mixed method study design.

DETAILED DESCRIPTION:
The Nigerian Agency for Food and Drug Administration and Control (NAFDAC) is leading implementation and scale-up of a national sodium reduction program with other national, state, and international agencies using the WHO's "Best Buy" SHAKE package (Surveillance of salt intake, Harness industry, Adopt standards for labelling and marketing, Knowledge to empower consumers, and Environments to promote healthy eating). SHAKE provides evidence-based recommendations for population-wide sodium reduction interventions for hypertension prevention and control.

The Nigeria Sodium Study will support this program's implementation and scale-up by evaluating the extent to which the program is implemented using a type III hybrid, mixed methods study design through repeated: 1) stakeholder interviews, 2) populations surveys, and 3) retail surveys. Implementation research methods will be used during adaptation, planning, and initial implementation for baseline (Wave 1) and follow-up Waves 2 and 3) assessments. A dietary sources of sodium study will also be performed at baseline and Wave 3 follow-up to target/track sodium reduction efforts according to local context and culture. Food retail surveys over the study period will capture novel data on packaged, unpackaged, and informal restaurant/hawker food through the international FoodSwitch program, which combines a consumer facing tool with crowdsourcing to better define Nigeria's food supply.

Investigators will use the Exploration, Preparation, Implementation and Sustainment (EPIS) framework throughout both phases. The formative research period will include Exploration and Preparation, when investigators will perform quantitative and qualitative measures of key process indicators, relevant contextual factors informed by CFIR, and relevant Proctor implementation outcomes, acceptability, feasibility and appropriateness. As implementation is started, investigators will use the Reach, Effectiveness, Adoption, Implementation and Maintenance (RE-AIM) framework, including implementation outcomes (feasibility, fidelity, adoption, acceptability, and cost) and contextual factors associated with the Implementation and Sustainment phases.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults (aged 18 to 69 years)
* Willingness to participate
* Permanent residents (a person who has been in the household for at least 6 months) of the study area
* Ability to provide informed consent

Exclusion Criteria:

* Individuals who are unable to provide informed consent
* Pregnant women, and those who are breastfeeding and/or women menstruating at the time of collection
* Cognitively impaired adults
* Those with known history of heart or kidney failure, stroke, liver disease
* Those who recently began therapy with diuretics (less than two weeks)
* Any other conditions that would make 24-hour urine collection difficult
* Individuals who are not yet adults (minors): i.e. infants, children, or teenagers <18 years old
* Prisoners or other detained individuals

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults will be enrolled as a single household representative from 3 states (Federal Capital Territory, Kano, and Ogun) of Nigeria.
Sampling Method: Probability Sample
Enrollment: 1350 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in mean population sodium intake from baseline (Wave 1) to follow-up (Waves 2 and 3). | Baseline (Wave 1) to follow-up (Wave 2 [estimated 18 months post-baseline] and Wave 3 [estimated 36 months post-baseline)
  Change in mean population sodium intake by age, sex, state, rurality, and presence of hypertension subgroups from baseline to Wave 2 and Wave 3 follow-up
Change in 24-hour urinary sodium from baseline (Wave 1) to follow-up (Wave 3) | Baseline (Wave 1) to follow-up (Wave 3 [estimated 36 months post-baseline)

SECONDARY OUTCOMES:
Change in overall and relative amount of dietary sources of sodium from baseline (Wave 1) to follow-up (Wave 3) | Baseline (Wave 1) to follow-up (Wave 3 [estimated 36 months post-baseline)
  Change in overall and relative amount of dietary sources of sodium (e.g., inherent in food, added during preparation, added at the table, added outside the home) by age, sex, state, rurality subgroups from baseline (Wave 1) to follow-up (Wave 3) based on the dietary sources of sodium study instruments.
Changes in self-reported knowledge, attitudes, and behavior about harms associated with excess sodium intake from baseline (Wave 1) to follow-up (Wave 3) | Baseline (Wave 1) to follow-up (Wave 3 [estimated 36 months post-baseline)
  Changes in self-reported knowledge, attitudes, and behavior about harms associated with excess sodium intake by age, sex, state, rurality subgroups from baseline (Wave 1) to follow-up (Wave 3) using based on the STEPS survey instrument.

OTHER OUTCOMES:
Change in mean population systolic and diastolic blood pressure from baseline (Wave 1) to follow-up (Waves 2 and 3). | Baseline (Wave 1) to follow-up (Wave 2 [estimated 18 months post-baseline] and Wave 3 [estimated 36 months post-baseline)
  Change in mean population systolic and diastolic blood pressure by age, sex, state, rurality subgroups.
Change in blood pressure lowering medication use | Baseline (Wave 1) to follow-up (Wave 2 [estimated 18 months post-baseline] and Wave 3 [estimated 36 months post-baseline)
  Change in blood pressure lowering medication use by age, sex, state, rurality subgroups.

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Huffman, MD, MPH, Principal Investigator — Washington University School of Medicine; Dike B Ojji, MD, PhD, Principal Investigator — University of Abuja Teaching Hospital
Locations (3):
- Nigeria (3):
  - Federal Medical Centre, Abeokuta, Ogun State
  - University of Abuja Teaching Hospital, Gwagwalada
  - Aminu Kano Teaching Hospital, Kano

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared through NHLBI BioLINCC.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available within 1 year of study conclusion.
Access Criteria: Access to study data will be managed through NHLBI BioLINCC